CLINICAL TRIAL: NCT01637779
Title: A Randomized Clinical Trial to Evaluate the Impact of a Fact Sheet About Childhood Immunization Pain Management on Parental Knowledge
Brief Title: A Randomized Controlled Trial About Teaching Parents How to Manage Childhood Immunization Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Anna Taddio, Associate Professor, Leslie Dan Faculty of Pharmacy, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 11-0231-E; 1000032989 (Other: The Hospital for Sick Children)
Record Dates: First submitted 2012-07-08; First posted 2012-07-11 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-10

CONDITIONS: Mothers of Newborn Infants
Keywords: randomized controlled trial; parent education; pain management; infant; immunization
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- fact sheet review (Experimental): mothers will review a fact sheet containing information about pain management during immunization then complete a knowledge test afterward
  Interventions: Behavioral: Fact sheet
- control unrelated material (Placebo Comparator): mothers will review material unrelated to pain management during immunization then complete a knowledge test
  Interventions: Behavioral: Fact sheet
- pre-test, review of fact sheet (Experimental): mothers do a pre-test, then read a fact sheet about how to manage immunization pain, then repeat the test
  Interventions: Behavioral: Fact sheet
- pre-test, control unrelated information (Placebo Comparator): mothers do a pre-test, then read unrelated material, then repeat the test
  Interventions: Behavioral: Fact sheet

INTERVENTIONS:
Behavioral: Fact sheet — fact sheet about pain management during immunization

SUMMARY:
There is no effect of a parent-directed fact sheet about pain management during childhood immunization and pre-test on parent learning about evidence-based pain relieving methods.

DETAILED DESCRIPTION:
Over 90% of young children demonstrate severe distress during vaccination. Pain relieving strategies are uncommonly used, despite a plethora of evidence for physical, pharmacological and psychological techniques. Parents commonly report pain as a harm-related concern for childhood immunizations and are dissatisfied with current practices. Unmitigated pain causes long-term adverse sequelae, including; anticipatory fear and hypersensitivity to pain at future procedures in children, and parental non-compliance with immunization schedules. Health providers and parents report the major barrier to routine use of pain management is parental lack of knowledge about effective strategies. Lack of time is reported as a secondary barrier. An educational tool about immunization pain management targeted to parents that can be practically implemented in the clinical setting within usual time constraints is needed.

ELIGIBILITY:
Inclusion Criteria:

* new mothers with health full-term infants
* 5 minute Apgar 7 or more

Exclusion Criteria:

* non-english speaking mothers
* mothers with psychiatric conditions
* infants admitted to intensive care unit

Ages: 15 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2012-07; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
knowledge | 10 minutes after intervention (educational material)
  maternal knowledge will be evaluated after reading the fact sheet or control (material unrelated to immunization)

SECONDARY OUTCOMES:
utilization of pain relieving interventions | 2 months after intervention
  maternal self-reported use of pain relieving interventions during routine 2-month infant immunizations

CONTACTS AND LOCATIONS:
Overall Officials: Anna Taddio, PhD, Principal Investigator — University of Toronto
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada